CLINICAL TRIAL: NCT04552418
Title: Pilot Study of Intestinal Microbiome Modification With Resistant Starch in Patients Treated With Dual Immune Checkpoint Inhibitors
Brief Title: Intestinal Microbiome Modification With Resistant Starch in Patients Treated With Dual Immune Checkpoint Inhibitors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMCC 2020.010; HUM00178229 (Other: University of Michigan)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor
Keywords: Immune checkpoint inhibitor
MeSH Terms: interventions — Resistant Starch

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Potato-based dietary starch supplement (Experimental): Patients undergoing cancer treatment with dual immune checkpoint inhibitors (ICI) will receive potato-based dietary starch supplements.
  Interventions: Drug: Potato starch

INTERVENTIONS:
Drug: Potato starch — Starting 5-7 days before treatment with dual-ICI, participant will consume 20g of potato starch (Bob's Red Mill®) once a day for 3 days, then increase to 20g twice a day, continuing throughout dual-ICI treatment (total duration approximately 13 weeks).
  Other Names: Resistant starch

SUMMARY:
This is a pilot study designed to assess the safety and feasibility of administering a dietary supplement to patients undergoing cancer treatment with a dual immune checkpoint inhibitors (ICIs) for solid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients starting dual immune checkpoint inhibitor therapy (ipilimumab and nivolumab in any dose combination) for solid cancer treatment per FDA approved indications.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with a history of colectomy and/or gastric bypass.
* Patients with a known diagnosis of inflammatory bowel disease or irritable bowel syndrome.
* Patients with active Clostridium difficile infection. Active infection is defined as a stool sample positive for Clostridium difficile toxin by EIA and either symptoms (frequent loose stools) OR imaging findings consistent with toxic megacolon.
* Inability to take oral supplements
* Patients with existing gastrointestinal symptoms including abdominal pain, diarrhea (watery stool), nausea and/or actively requiring regular anti-emetics.
* Patients with symptomatic bowel metastasis including pain, severe constipation, or gastrointestinal bleeding.
* Receiving antibiotic within 14 days of ICI therapy initiation.
* Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient or raise concern that the patient would not comply with protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Number of patients able to adhere to resistant starch (RS) supplement schedule | Approximately 13 weeks
  Feasibility will be determined by calculating the number of patients who have taken 70% or more of scheduled dose of dietary intervention. Patients will be asked to record doses of starch taken and will be provided a table in which doses can be checked off.
Frequency of serious adverse events (SAEs) attributable to ICI therapy | Up to 6 months (3 months after RS supplement discontinuation)
  Adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency of known serious effects of ICIs will be compared to historical rates.
Occurrence of unanticipated serious adverse events (SAEs) | Approximately 13 weeks
  Adverse events will be assessed using the NCI CTCAE, version 5.0.

SECONDARY OUTCOMES:
Incidence and severity of immunotherapy-induced diarrhea/colitis | Up to 6 months (3 months after RS supplement discontinuation)
  Graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Change in luminal microbiome composition | Up to 6 months (3 months after RS supplement discontinuation)
  Weekly stool samples will be compared to the baseline sample (prior to starting starch-based dietary supplement). Stool samples will be analyzed for microbial nucleic acids to characterize the components of the stool microbiome.
Change in luminal microbiome metabolite | Up to 6 months (3 months after RS supplement discontinuation)
  Weekly stool samples will be compared to the baseline sample (prior to starting starch-based dietary supplement). Key metabolic byproducts will be identified in stool specimens using liquid chromatography and mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Fecher, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No